CLINICAL TRIAL: NCT01324648
Title: A Randomized Controlled Trial Evaluation of Brief, Telephone Supported CBT Self-help in Primary Care Patients With Mild to Moderate Depression
Brief Title: Evaluation of the Bounce Back Program
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Canadian Mental Health Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H08-02847; 106504 (Other Grant/Funding Number: Canadian Institute of Health Research)
Record Dates: First submitted 2011-03-14; First posted 2011-03-29 (Estimated); Last update posted 2014-09-10 (Estimated); Status verified 2014-09

CONDITIONS: Depression
Keywords: Guided self-help; Telephone delivery; Cognitive behavior therapy; Bibliotherapy
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- TG + GP TAU (Experimental)
  Interventions: Behavioral: Telephone-supported self-help and GP treatment as usual
- UG + GP TAU (Experimental)
  Interventions: Behavioral: Unsupported self-help and GP treatment as usual
- GP TAU (Active Comparator)
  Interventions: Other: General practitioner treatment as usual

INTERVENTIONS:
Behavioral: Telephone-supported self-help and GP treatment as usual — Participants' use of the BB self-help materials will be supported by three to five telephone coaching sessions that occur approximately every 2-3 weeks. Total contact time will be approximately 2 hours (2 hour total contact time will be considered "brief" in our study). Participants will also continue to receive whatever current treatment their general practitioner is providing.
  Arms: TG + GP TAU
Behavioral: Unsupported self-help and GP treatment as usual — This treatment was chosen as a control for the telephone coaching component of the BB program. Participants will be sent a package containing the BB self-help materials and along with instructions on how to utilize these materials. Participants will use the materials on their own and at their own pace. Participants will also continue to receive whatever current treatment their general practitioner is providing.
  Arms: UG + GP TAU
Other: General practitioner treatment as usual — This group will receive treatment as usual - whereby the clinic staff will inform the participant's GP of their PHQ-9 score. They will also be informed that their GP will be contacted that they are taking part in the research and that their GP will continue to support them with their depression as usual.
  Arms: GP TAU

SUMMARY:
Lifetime prevalence rates of Major Depressive Disorder (MDD) in Canada are between 10-12% with approximately 1.5 million Canadians reporting depression in any given year. Alarmingly, the burden of ill health associated with MDD is projected to increase worldwide such that by the year 2020, depression will move from its current position of fourth to become the second greatest burden of ill health, closely following ischaemic heart disease (Murray & Lopez, 1998). As depressed patients are often in frequent contact with their primary care physicians for other health problems, effective depression treatment and management currently relies heavily on the primary care sector. Cognitive behavioural therapy (CBT) is an empirically supported psychotherapy that is recommended by the Canadian Network for Mood and Anxiety Treatments Clinical Guidelines as a first-line treatment for depression. However, across Canada, CBT is not readily accessible by primary care physicians for their patients, particularly in rural areas.

To help address this nationwide need for CBT, British Columbia (BC) is the first and only province in Canada to develop and implement a high capacity mental health service, Bounce Back: Reclaim your Health (BB), for primary care patients with mild to moderate depression. In BB, the patients' use of Cognitive-Behavioural Therapy (CBT) self-help materials is supported via trained telephone coaches.

The primary objective of our proposed research is to provide direct evidence of the effectiveness of the BB program, and, in particular, the telephone coaching component. The investigators will test: (1) whether the BB program is more effective than general practitioner (GP) treatment-as-usual (TAU); and (2) whether BB's positive results can be attributed to the telephone coaching component, as this component is associated with the most significant costs of the program. A secondary objective is to assess the cost-effectiveness of such telephone support.

DETAILED DESCRIPTION:
This proposed project is designed to evaluate and provide direct evidence for the clinical effectiveness of the Bounce Back: Reclaim your Health (BB) project currently implemented in 17 communities in British Columbia (BC). BB is an innovative mental health service in the health care system designed to help patients participate in their own care by teaching them the sufficient and necessary skills to manage their moods. This BB program, led by the Canadian Mental Health Association's BC Division, offers mental health support to primary care patients suffering from mild to moderate depression. BB is a low intensity, high capacity program, based on cognitive behaviour therapy (CBT) self-help materials Overcoming Depression, Low Mood and Anxiety: A five areas approach (OD - comprising psycho-educational DVD and self-help mood improvement workbook). The content of these self-help materials was adapted to a BC context for the BB program. In addition, in order to best meet the needs of BC primary care patients, this new mental health service is delivered to patients in their own homes and patients' use of the OD self-help materials is supported via trained telephone coaches. Telephone coaches are non-specialists trained and monitored by a registered psychologist. Coaching enables patients to engage with and get the most out of the materials. The advantages of telephone coaching include privacy, accessibility, and convenience, especially for those patients living in rural areas and can not access treatment due to geographic barriers; those who do not seek treatment due to stigma; or those who are coping with chronic physical illness and multiple medical appointments. There is only indirect support for the effectiveness of the BB program. Thus, this proposed project is designed to evaluate and provide direct evidence of the effectiveness of the BB program.

ELIGIBILITY:
Inclusion Criteria:

* currently experiencing a mild to moderate level of depressive symptoms as defined by a score of 5 - 19 on the PHQ-9;
* 19 years of age or older
* willing to use the BB program;
* able to use the BB self-help materials with telephone coaching (have access to read, hear a telephone conversation and have a telephone); and,
* ability to give informed consent and complete questionnaires unassisted.

Exclusion Criteria:

* a SCID diagnosis (past or present) of: (a) Bipolar Disorder; (b) Schizophreniform Disorders; (c) Substance Abuse or Dependence (current or within the past six months); (d) Borderline or Antisocial Personality Disorder (based on GP's diagnosis); or (e) Cognitive Disorder (as the BB program is not appropriate for these individuals);
* active suicidal intent, (as defined by a score of 2 or more on the BDI-II suicide item #9; those with passive suicidal ideation will be monitored;
* impaired concentration and motivation (scoring 7 or more on the combined BDI-II items #15, 19 and 20 for energy, concentration difficulty and tiredness, respectively);
* are currently receiving, or have received in the previous 6 months, CBT or guided self-help for depression; or,
* are involved in other clinical research studies.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Estimated)
Dates: Start 2011-03; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Changes in levels of depressive symptomatology | The PHQ-9 will be assessed at screening, 2 month, 4 month, and 12 month time points.
  Levels of depressive symptomatology will be measured over time, using the Patient Health Questionnaire (PHQ-9)

SECONDARY OUTCOMES:
Changes of levels of anxiety | The GAD-7 will be assessed at baseline, 2 month, 4 month, and 12 month time points
  Levels of anxiety will be measured over tiem, using the Generalized Anxiety Disorder 7 (GAD-7).
Changes in quality of life and enjoyment | The QLES-Q-SF will be assessed at baseline, 2 month, 4 month, and 12 month time points
  Quality of life and enjoyment will be measured over time using the Quality of Life and Enjoyment Satisfaction Questionnaire (QLES-Q-SF).
Changes in work and social adjustment | The WASA will be assessed at baseline, 2 month, 4 month, and 12 month time points
  Work and social adjustemnt will be assessed over time, using the Work and Social Adjustment Scale (WASA).
Changes in work functionality and impairment | The LEAPS will be assessed at baseline, 2 month, 4 month, and 12 month time points
  Work functionality and impairment will be assessed over time using the Lam Employment and Productivity Scale (LEAPS).
Changes in mental health literacy | The MHL-Q will be assessed at baseline, 2 month, 4 month, and 12 month time points
  Mental health literacy will be measured over time using the Mental Health Literacy questionnaire (MHL-Q).
Changes in use of health services | The CSRI will be asssessed at screening, 4 month, and 12 month time points
  Participants' use of health services will be assessed using the Client Service Receipt Inventory - modified (CSRI).
Changes in health status | The EQ-5D will be assessed at baseline, 2 month, 4 month, and 12 month time points
  Health status will be assessed using the Euroquol-5 (EQ-5D).
Changes in health status and health related quality of life | The HUI-3 will be assesed at baseline, 2 month, 4 month, and 12 month time points
  Health status and health related quality of life will be assessed over time using the Health Utilities Index (HUI-3).
Changes in illness severity | The DUSOI will be assessed at baseline, 2 month, 4 month, and 12 month time points
  Illness severity will be assessed over time using the Duke Severity of Illness Checklist (DUSOI).
Client satisfaction. | The CSQ-9 will be assessed at 4 month time point.
  Client satisfaction will be assessed using the Client Satisfaction Questionnaire 9 (CSQ-9).

CONTACTS AND LOCATIONS:
Overall Officials: Mark Lau, PhD, Principal Investigator — University of British Columbia
Locations (3):
- Canada (3):
  - Calgary Foothills Primary Care Network, Calgary, Alberta
  - Chinook Primary Care Network, Chinook Valley, Alberta
  - University of British Columbia, Vancouver, British Columbia

REFERENCES:
- See also: Related Info — http://www.cmha.bc.ca/bounceback